CLINICAL TRIAL: NCT01528137
Title: A Phase Ib Immunomodulatory Study of Single Agent Talactoferrin in Patients With Select Relapsed or Refractory Non-Small Cell Lung Cancer (NSCLC) and Squamous Head and Neck Cancer (HNSCC)
Brief Title: Talactoferrin in Treating Patients With Relapsed or Refractory Non-Small Cell Lung Cancer or Squamous Cell Head and Neck Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Negative data from another trial led to termination of this trial by sponsor.
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Agennix (Industry)
Responsible Party: Principal Investigator, Heather Wakelee, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAR0072; NCI-2012-00060 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23170 (Other: Stanford University IRB)
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Salivary Gland Squamous Cell Carcinoma; Stage III Salivary Gland Cancer; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Non-small Cell Lung Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IVA Salivary Gland Cancer; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Salivary Gland Cancer; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Salivary Gland Cancer; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Verrucous Carcinoma of the Larynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Tongue Neoplasms | interventions — talactoferrin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (immunomodulator) (Experimental): Patients receive talactoferrin PO BID for 12 weeks. Courses repeat every 14 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: talactoferrin; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: talactoferrin — Given PO
  Other Names: oral recombinant human lactoferrin; oral rhLF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies how well talactoferrin works in treating patients with relapsed or refractory non-small cell lung cancer (NSCLC) or squamous cell head and neck cancer. Biological therapies, such as talactoferrin, may stimulate the immune system in different ways and stop tumor cells from growing

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Monitoring of immunologic response to therapy in tumor tissue and peripheral blood. Identification of potential candidate biomarkers indicating clinical benefit to talactoferrin.

SECONDARY OBJECTIVES:

I. Progression free survival (PFS), objective response rate (ORR), stable disease (SD), overall survival (OS), disease stability, and disease stability at 7 weeks.

OUTLINE:

Patients receive talactoferrin orally (PO) twice daily (BID) for 12 weeks. Courses repeat every 14 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up monthly for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed, incurable metastatic relapsed/refractory NSCLC or relapsed/refractory, incurable, locally advanced or metastatic squamous head and neck cancer Head and neck squamous cell cancer patients must be able to be biopsied safely in clinic or by Stanford Interventional Radiology as determined by a Stanford Head and Neck Oncologist or Stanford Head and Neck Surgeon Hemoglobin (Hgb) >= 9 gm/dl Platelets >= 80,000/uL International normalized ratio (INR) =< 1.5 Total bilirubin =< 1.5 Creatinine =< 1.5 Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2 times the upper limit of normal Failed therapy with at least one standard first line chemotherapy regimen, or intolerant of standard chemotherapy At least 4 weeks from the last chemotherapy, immunosuppressive/immunomodulatory therapy or investigational agent and 2 weeks from erlotinib or other non-immunogenic therapy Palliative radiotherapy to painful bony metastases must be completed at least 2 weeks prior to initiation of study treatment Brain metastases must be adequately treated (stable and asymptomatic) with surgery and/or radiation prior to enrollment and any steroids completed at least 3 weeks prior to study treatment initiation At least one un-irradiated target lesion measurable by Response Evaluation Criteria In Solid Tumors (RECIST) criteria At least one lesion amenable to repeat biopsy Life expectancy of at least 2 months Eastern Cooperative Oncology Group (ECOG) performance status 0-2 Absolute neutrophil count >= 1,000/µl Absolute lymphocyte count >= 800/µl Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

Concomitant chemotherapy, radiotherapy, immunosuppressive/immunomodulatory therapy or investigational agents Head and Neck Squamous Cell Carcinoma that can not be safely biopsied in Head and Neck Oncology Clinic or by Stanford Interventional Radiology as determined by a Stanford Head and Neck Oncologist or a Stanford Head and Neck Surgeon

Co-morbid disease or incurrent illness that could affect patients' immune status or ability to comply with the study, but not limited to:

* Renal failure requiring hemodialysis;
* New York Heart Association (NYHA) Grade III or greater congestive heart failure;
* Unstable angina;
* Severe infectious or inflammatory illness;
* Human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS);
* Hepatitis (Hep) C positive (+) or Hep B surface antigen (+) Second malignancy with less than 5 years since documented clinical remission except for non-melanoma skin cancers or curatively treated cervical carcinoma in situ, superficial bladder cancer or early prostate cancer Prior history of allergic reaction to compounds of similar chemical or biologic composition to talactoferrin Inability to comply with study and/or follow-up procedures because of psychiatric or social situations Pregnant and nursing patients, sexually active patients (male and female) unwilling to practice contraception while on the study and at least 30 days after completion Oral corticosteroid therapy within 2 weeks prior to randomization or expected to be ongoing during the study Any gastrointestinal tract disease or other medical condition resulting in the inability to take oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Correlation of changes in cytokine composition and other immunologic measurements in tumor, tumor stroma and blood with benefit to talactoferrin | Baseline and weeks 2, 7, 14, 21, and 49
  Descriptive statistics and trends in cytokine and immunological parameters both in the tumor biopsies and the blood samples will be summarized.

SECONDARY OUTCOMES:
PFS | Duration of time from start of treatment to time of documented progression or death up to at least 12 months
ORR | Baseline and then every 7 weeks
SD | Baseline and then every 7 weeks
OS | Time from the date of enrollment to the date of death due to any cause or the last date the patient was known to be alive (censored observation) at the date of data cutoff for the final analysis up to at least 12 months
Disease stability | Baseline and then every 7 weeks
Disease stability | At 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Heather Wakelee, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States